CLINICAL TRIAL: NCT02269670
Title: Phase II Study of Everolimus Beyond Progression in Postmenopausal Women With Advanced, Hormone Receptor Positive Breast Cancer
Brief Title: Phase II Study of Everolimus Beyond Progression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow to accrual
Sponsor: Emory University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Suchita Pakkala, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00071229; NCI-2014-02092 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); WINSHIP2563-13 (Other: Emory University/Winship Cancer Institute)
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Results first posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Estrogen Receptor-positive Breast Cancer; HER2-negative Breast Cancer; Progesterone Receptor-positive Breast Cancer; Recurrent Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; Anastrozole; Letrozole; Tamoxifen; Fulvestrant; Megestrol Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (everolimus, hormone therapy) (Experimental): Patients receive everolimus PO daily and a hormone therapy regimen chosen at the discretion of the investigator (anastrozole PO daily; letrozole PO daily; tamoxifen citrate PO daily; fulvestrant IM or PO on days 1, 15, and 29, and then monthly; megestrol acetate PO QID; or other regimen). Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: everolimus; Drug: anastrozole; Drug: letrozole; Drug: tamoxifen citrate; Drug: fulvestrant; Drug: megestrol acetate

INTERVENTIONS:
Drug: everolimus — Given PO
  Other Names: 42-O-(2-hydroxy)ethyl rapamycin; Afinitor; RAD001
Drug: anastrozole — Given PO
  Other Names: ANAS; Arimidex; ICI-D1033
Drug: letrozole — Given PO
  Other Names: CGS 20267; Femara; LTZ
Drug: tamoxifen citrate — Given PO
  Other Names: Nolvadex; TAM; tamoxifen; TMX
Drug: fulvestrant — Given IM or PO
  Other Names: Faslodex; ICI 182,780
Drug: megestrol acetate — Given PO
  Other Names: BDH 1298; Maygace; Megace; Megestil; Niagestin

SUMMARY:
This phase II trial studies how well everolimus and hormone therapy work in treating patients with hormone receptor positive breast cancer that has continued to spread (progressed) or returned after a period of improvement (recurred) on everolimus and exemestane hormone therapy. Everolimus is a chemotherapy drug that may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Estrogen and progesterone are hormones that can cause the growth of breast cancer cells. Hormone therapy may fight breast cancer by lowering the amount of estrogen and progesterone the body makes. Giving everolimus with a different type of hormone therapy may be an effective treatment for breast cancer in patients who progressed on everolimus with exemestane.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

Progression free survival in patients with advanced or metastatic breast cancer receiving everolimus plus hormonal therapy beyond first progression.

SECONDARY OBJECTIVES:

1. Clinical benefit rate (sum of stable disease, partial response, complete response).
2. Response rate (partial response and complete response).
3. Overall survival.
4. Safety, side effects and tolerability profile of everolimus.

OUTLINE:

Patients receive everolimus orally (PO) daily and a hormone therapy regimen chosen at the discretion of the investigator (anastrozole PO daily; letrozole PO daily; tamoxifen citrate PO daily; fulvestrant intramuscularly [IM] or PO on days 1, 15, and 29, and then monthly; megestrol acetate PO 4 times daily [QID]; or other regimen). Treatment continues in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Estrogen (ER) and/or progesterone (PR)-positive at primary diagnosis and at metastatic diagnosis where tissue is available (defined as > or = 1% of staining nuclei)
* Progressive or recurrent breast cancer defined as disease progression or recurrence while on a combination of exemestane with everolimus
* Human epidermal growth factor receptor 2 (HER2)/neu-negative breast cancer by standard criteria (immunohistochemistry [IHC] < 3+ or fluorescence in situ hybridization [FISH] negative if IHC 2+) at primary diagnosis
* Histologically confirmed, measurable or evaluable disease; patients should have at least one measurable lesion; if applicable, Response Evaluation Criteria in Solid Tumors (RECIST) criteria should be used
* Life expectancy > 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Absolute neutrophil count (ANC) > 1,500/µL
* Platelets ≥ 100,000/µL
* Hemoglobin > 10 g/dL
* Creatinine ≤ 1.5 x upper limit of normal (ULN)
* Bilirubin ≤ 1.5 x ULN
* International normalized ratio ≤ 1.3 (or ≤ 3 on anticoagulants)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2 x ULN unless related to primary disease
* Signed informed consent
* Adequate birth control
* Fasting serum cholesterol ≤ 300 mg/dL OR ≤ 7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN; NOTE: in case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication

Exclusion Criteria:

* Prior treatment with everolimus other than in combination with hormonal therapy for treatment of breast cancer or prior treatment with another mammalian target of rapamycin (mTOR) inhibitor (sirolimus, temsirolimus) for any indication
* HER2 positive disease as defined by 3+ IHC or positive FISH (both in primary and metastatic sites)
* Active infection: temperature > 100 Fahrenheit (F), fever of unknown origin, active symptoms or signs of infection as defined by the investigator
* Uncontrolled central nervous system metastases
* Life-threatening, visceral metastases
* Pregnant or lactating women
* Prior chemotherapy within the last 4 weeks
* Prior radiation therapy within the last 4 weeks; prior radiation therapy to indicator lesion (unless objective disease recurrence or progression within the radiation portal has been documented since completion of radiation)
* Concomitant malignancies or previous malignancies within the last 5 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* History of significant cardiac disease, cardiac risk factors or uncontrolled arrhythmias
* Hypersensitivity to trial medications (everolimus)
* Emotional limitations, which the investigator judges could limit the patient's ability to follow up and comply with study procedures
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent
* Uncontrolled diabetes as defined by fasting serum glucose > 1.5 x ULN
* Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* A known history of human immunodeficiency virus (HIV) seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of EVEROLIMUS (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active, bleeding diathesis
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods; if barrier contraceptives are being used, these must be continued throughout the trial by both sexes; hormonal contraceptives are not acceptable as a sole method of contraception; (women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of EVEROLIMUS)
* Symptomatic intrinsic lung disease or extensive tumor involvement of the lungs, resulting in dyspnea at rest
* Taking any of the following agents:

  * Chronic treatment with systemic steroids or another immunosuppressive agent (use of steroids as part of management of everolimus toxicities will be allowed)
  * Live vaccines
  * Patients who have received live attenuated vaccines within 1 week of start of everolimus and during the study; patient should also avoid close contact with others who have received live attenuated vaccines; examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, bacillus Calmette-Guérin (BCG), yellow fever, varicella and TY21a typhoid vaccines
  * Drugs or substances known to be inhibitors or inducers of the isoenzyme cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A)

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-11-25 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suchita Pakkala, MD, Principal Investigator — Emory University/Winship Cancer Institute
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Everolimus, Hormone Therapy)
Started | 3
Completed | 0
Not Completed | 3
Not completed — All subjects have not completed all research related interventions | 3

BASELINE CHARACTERISTICS:
Population: No data displayed because Outcome Measure has zero total analyzed.
Arm/Group | Treatment (Everolimus, Hormone Therapy)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Partial Response Plus Complete Response) Using RECIST
Description: Study was terminated early due to difficulties with enrollment. No outcome measures were assessed.
Time Frame: Up to 2 years
Population: Study was terminated early due to difficulties with enrollment. No outcome measures were assessed.
Arm/Group | Treatment (Everolimus, Hormone Therapy)
Number analyzed (Participants) | 0

2. Primary Outcome: Progression-free Survival (PFS)
Description: Study was terminated early due to difficulties with enrollment. No outcome measures were assessed.
Time Frame: Up to 2 years
Population: Study was terminated early due to difficulties with enrollment. No outcome measures were assessed.
Arm/Group | Treatment (Everolimus, Hormone Therapy)
Number analyzed (Participants) | 0

3. Secondary Outcome: Clinical Benefit Rate (Response Rate Plus Stable Disease)
Description: Study was terminated early due to difficulties with enrollment. No outcome measures were assessed.
Time Frame: Up to 2 years
Population: Study was terminated early due to difficulties with enrollment. No outcome measures were assessed.
Arm/Group | Treatment (Everolimus, Hormone Therapy)
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival (OS)
Description: Study was terminated early due to difficulties with enrollment. No outcome measures were assessed.
Time Frame: From the initiation of alternate hormonal treatment in combination with everolimus to time of death from any cause, assessed up to 2 years
Population: Study was terminated early due to difficulties with enrollment. No outcome measures were assessed.
Arm/Group | Treatment (Everolimus, Hormone Therapy)
Number analyzed (Participants) | 0

5. Secondary Outcome: Incidence of Adverse Events Assessed Using Common Terminology Criteria for Adverse Events Version 4.0
Description: Study was terminated early due to difficulties with enrollment. No outcome measures were assessed.
Time Frame: Up to 2 years
Population: Study was terminated early due to difficulties with enrollment. No outcome measures were assessed.
Arm/Group | Treatment (Everolimus, Hormone Therapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year
Arm/Group | Treatment (Everolimus, Hormone Therapy)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Everolimus, Hormone Therapy) (N=3)
Hypothyroidism (Endocrine disorders) | 1 (1)
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Metabolism and nutrition disorders) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2)
Creatinine increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (2)

LIMITATIONS AND CAVEATS:
Early termination of the study because of recruitment difficulties lead to insufficient data collection and analysis of primary and secondary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-12-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT02269670/Prot_001.pdf
  • Informed Consent Form (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/70/NCT02269670/ICF_000.pdf